CLINICAL TRIAL: NCT03876782
Title: Level of Agreement of Intraocular Lens Power Measurements Between IOLMaster and Verion
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: Th9/ES2/22-2-19
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Cataract
Keywords: cataract surgery; Verion Image-Guided System; IOLMaster; IOL calculation; keratometry; corneal power; toric IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IOLMaster group: IOL power for all cataract participants will be measured with IOLMaster and Verion
  Interventions: Diagnostic Test: IOLMaster; Diagnostic Test: Verion

INTERVENTIONS:
Diagnostic Test: IOLMaster — IOL power calculation will be done with IOLMaster
Diagnostic Test: Verion — IOL power calculation will be done with Verion

SUMMARY:
Primary objective of this study is to evaluate the level of agreement of two keratometry modules, the IOLMaster and the Verion Reference Unit, in terms of keratometric values and IOL power calculation.

DETAILED DESCRIPTION:
Participants were enrolled from the Cataract & Presbyopia Service of the University General Hospital of Alexandroupolis in a consecutive-if-eligible basis. Apart from keratometric values, IOL power calculations will be compared for 8 IOL models (Acrysof SN60WF, SN60AT, SN6ATx, TFNT00, TFNTx0, SV25T0, SV25Tx and Tecnis ZCB00) using 4 formulas (SRK/T, Holladay 1, Hoffer Q and Haigis).

ELIGIBILITY:
Inclusion Criteria:

* Senile Cataract

Exclusion Criteria:

* Former incisional surgery,
* Corneal diseases,
* Dry-eye-Disease,
* Glaucoma drops,
* Inability to obtain accurate measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract patient that visit the Cataract Outpatients Service of the University Hospital of Alecxnadroupolis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
IOL Power Calculation | 1 day prior to surgery
  Exact calculation of dioptric power of the intraocular lens

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Associate Professor
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece